CLINICAL TRIAL: NCT00519402
Title: Outcomes of Partial Versus Complete Tonsillectomy for Obstructive Sleep Disordered Breathing in Children
Brief Title: Outcomes of Partial Versus Complete Tonsillectomy for Obstructive Sleep Disordered Breathing
Status: Withdrawn | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, michael macknin, Staff, General Pediatrics, The Cleveland Clinic
Other Study IDs: 07-433
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Disordered Breathing
Keywords: partial tonsillectomy; complete tonsillectomy; tonsillectomy; obstruction sleep disordered breathing OSDB; apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Partial Tonsillectomy: Patients who received a partial tonsillectomy
  Interventions: Other: tonsillar examination and questionnaire completion
- Complete Tonsillectomy: Patients who received a complete tonsillectomy
  Interventions: Other: tonsillar examination and questionnaire completion

INTERVENTIONS:
Other: tonsillar examination and questionnaire completion

SUMMARY:
Introduction: There is currently no long-term study, which compares the outcomes of partial tonsillectomy to conventional tonsillectomy. We hypothesize that there will be little significant tonsillar regrowth with partial tonsillectomy.

Background and Significance: Tonsillectomy is the most common major surgical procedure performed on children in the United States with nearly 300,000 procedures performed each year, primarily for the indication of obstructive sleep disordered breathing (OSDB). Conventional (total) tonsillectomy removes the tonsillar capsule, and partial tonsillectomy preserves the capsule by shaving away the tonsils using an endoscopic microdebrider. Partial tonsillectomy results in less pain, fewer days to normal activity and diet, and fewer days of analgesics than total tonsillectomy. There are no significant differences between the techniques in blood loss or postoperative life improved Historical evidence suggests that eventually there will be tonsillar regrowth with partial tonsillectomy. However, in a 2003 follow-up report of 243 children undergoing partial tonsillectomy and 107 undergoing complete tonsillectomy from 1998 through 2002 for OSDB there was no evidence of significant tonsillar regrowth. (1) We will follow-up children undergoing partial or complete tonsillectomies at the Cleveland Clinic from 1998 through 2002. There will be standardized tonsillar examinations by two observers, with a third observer in cases of significant disagreement, and questionnaires evaluating sleep apnea and daytime sleepiness, and number of tonsillar infections.

If there are a large number of children with recurrent tonsillar symptoms post partial tonsillectomy, the procedure should be abandoned. However, if follow-up reveals comparable tonsillar symptoms for partial and the total tonsillectomy, perhaps the partial procedure should replace the total tonsillectomy as the standard operation to relieve tonsillar OSDB. This could eventually result in millions of less lost days of work and school in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing tonsillectomies at the Cleveland Clinic from 1998-2002

Ages: 5 Years to 28 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing tonsillectomies at the Cleveland Clinic from 1998-2002
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Macknin, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States